CLINICAL TRIAL: NCT03245931
Title: Hepatitis C Education for Pregnant Women With Opiate Addiction - Phase 1
Status: Completed | Type: Observational
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 17007
Record Dates: First submitted 2017-07-21; First posted 2017-08-10 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Qualitative Interview — Complete 6 open-ended qualitative questions on patients in the HOPE program to assess basic current understanding about Hepatitis C and topics of interest that patients in the HOPE program would like to learn more about.

SUMMARY:
The goal of this study is to assess the health literacy level of patients enrolled in the HOPE program, identify any gaps in their knowledge of hepatitis C, analyze the variables that may influence patients' knowledge, and educate patients on Hepatitis C.

DETAILED DESCRIPTION:
The study will compare the effectiveness of providing a pamphlet and expert education compared to providing a pamphlet only. The information gained in completing this study will help the medical community improve patient education on the disease and specifically understand how the medical community can best serve pregnant patients with opiate dependence burdened by Hepatitis C.

ELIGIBILITY:
Inclusion Criteria

* The study will include patients with and without Hepatitis C diagnosis.
* Patients will be recruited at their routine prenatal and post-partum visits.
* Patients who speak and understand English

Exclusion Criteria:

* Patients under the age of the 18 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population includes obstetrics patients enrolled in the HOPE program who are 18 years old or older.
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2019-08-26 (Actual)

PRIMARY OUTCOMES:
Discovering the gaps in patients' knowledge of Hepatitis C | 2 months
  Through interview, 6 open-ended qualitative questions will be asked of the patients in the HOPE program to assess basic current understanding about Hepatitis C

CONTACTS AND LOCATIONS:
Overall Officials: Michael Marcotte, MD, Principal Investigator — TriHealth Inc.
Locations (1):
- Good Samaritan Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No